CLINICAL TRIAL: NCT06024148
Title: Evaluation of the Continuation of Anti-osteoporotic Treatment 1 Year After Initial Administration Following Severe Osteoporotic Fracture in Patients Aged 75 and Over, Hospitalized at the Rocheplane Medical Center
Brief Title: Continuation of Anti-osteoporotic Treatment 1 Year After Initial Administration
Acronym: POUROSTEO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0179
Record Dates: First submitted 2023-08-17; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Osteoporosis Fracture
Keywords: antiosteoporotic treatment; professional practice assessment
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients hospitalized in the Geriatric Rehabilitation Department: patients aged 75 and over, admitted with a severe osteoporotic post-fracture, having received a first dose of antiosteoporotic treatment between the day of fracture and discharge from Geriatric Rehabilitation Department
  Interventions: Other: phone survey

INTERVENTIONS:
Other: phone survey — patients complete a 10-minute telephone questionnaire on their osteoporosis management

SUMMARY:
The aim of this observational study is to assess the obstacles and levers to the continuation of anti-osteoporotic treatment, and to identify those where action could be taken to improve the quality of care for fractured patients.

The individual and collective stakes are high. Fracture is the most feared complication of osteoporosis. The current under-diagnosis and under-treatment of this chronic pathology exposes patients to a high risk of early re-fracture, with the associated morbidity and mortality.

General practitioners have a major role to play in monitoring and coordinating patients' healthcare pathways. The aim of this study is to assess ways of improving osteoporosis management in order to improve quality of life and disability-free life expectancy for individual patients. The public health and economic stakes are equally high. It is by identifying the obstacles that prospective work on the key elements to be implemented could help optimize osteoporosis management.

DETAILED DESCRIPTION:
Selection of patients hospitalized at the Rocheplane Medical Center between June 2021 and May 2022, following a severe osteoporotic fracture and having received a first dose of antiosteoporotic treatment during their overall stay (initial admission department + CMR).

Sending of an information letter and request for non-objection from patients or their trusted support person, with a 1-month cooling-off period to express opposition.

Collection of variables of interest from CMR patients' medical records, followed by administration of a telephone hetero-questionnaire (transferred to Excel) to patients or their families 1 year after fracture occurrence.

If the patient or family did not answer the questionnaire, or if it was incomplete (missing data), the information could be sought by telephone from the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in CMR's Geriatric Rehabilitation Department between 01/06/2021 and 31/05/2022
* Age: 75 and over
* Admitted with severe post-fracture osteoporosis
* Having received a first dose of antiosteoporotic treatment between the day the fracture occurred and discharge from CMR (either in an inpatient unit prior to CMR, or at CMR)

Exclusion Criteria:

* Having objected to the use of his/her data for research purposes
* Subject under guardianship or deprived of liberty.
* Pathological fracture
* Anti-osteoporotic treatment prior to fracture
* 1-year follow-up made impossible by lack of contact with patient, family or attending physician.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will include the number of patients corresponding to the "patient flow" admitted to CMR's units of interest over one year, and, corresponding to the inclusion criteria (CMR welcomes 250 patients aged 75 and over to its geriatric units each year, all types of fractures combined; ¾ of patients are admitted for severe fractures).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of continuation of anti-osteoporotic treatment at 1 year after initial administration following a severe osteoporotic fracture in patients aged 75 and over. | Telephone data collection one year after Geriatric Rehabilitation Department stay
  Percentage of patients for whom anti-osteoporosis treatment was renewed 1 year after initial administration (between fracture occurrence and discharge from the geriatric department)

SECONDARY OUTCOMES:
Determine the rate of introduction of anti-osteoporotic treatment during the patient's overall stay | Medical records collected one year after Geriatric Rehabilitation Department stay
  Percentage of patients who received anti-osteoporosis treatment during their overall stay
Identify patient-related obstacles and levers to treatment renewal at 1 year after fracture | Telephone data collection one year after Geriatric Rehabilitation Department stay
  Percentage of patients presenting: a contraindication to treatment, intolerance to treatment, refusal of treatment, non-adherence to treatment, failure to consult their GP, forgetfulness, death.
Determine the obstacles and levers to the continuation of treatment at 1 year after a fracture, in relation to the treating physician. | Telephone data collection one year after Geriatric Rehabilitation Department stay
  Percentage of GPs reporting: unfamiliarity with the introduction of treatment at the time of fracture, unfamiliarity with how to prescribe treatment, unfamiliarity with "osteoporosis" recommendations, non-prescribing for fear of adverse effects (iatrogenicity), non-prescribing based on a judgement of an unfavourable benefit/risk balance, feeling of incompetence regarding the management of osteoporosis, lack of time, proposing therapeutic alternatives, forgetfulness.
Determine the obstacles and levers to the continuation of treatment at 1 year for fractures related to the healthcare system | Telephone data collection one year after Geriatric Rehabilitation Department stay
  Absence of clear follow-up instructions on upstream department reports (quality of inter-professional communication), Absence of consultation with a rheumatologist, Absence of consultation with a geriatrician, Difficulty accessing a dental consultation, Absence of BMD, Cost of medication, Existence of a doctor-pharmacist link, GP cooperation with a network of well-identified specialists.
Evaluation of the professional practices of general practitioners concerning the management of osteoporosis. | Telephone data collection one year after Geriatric Rehabilitation Department stay of their patient
  Analysis of the results of the professional practice assessment questionnaire